CLINICAL TRIAL: NCT02965703
Title: Evaluating Intermittent Dosing of Aspirin for Colorectal Cancer Chemoprevention
Brief Title: Aspirin in Preventing Colorectal Cancer in Patients With Colorectal Adenoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2016-01642; NCI-2016-01642 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; NCI2015-06-01 (Other: Northwestern University); NWU2015-06-01 (Other: DCP); N01CN00035 (NIH); P30CA060553 (NIH)
Record Dates: First submitted 2016-11-16; First posted 2016-11-17 (Estimated); Results first posted 2025-03-04 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Adenoma; Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin; Specimen Handling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (aspirin) (Experimental): Patients receive aspirin PO daily for 12 weeks in the absence of unacceptable toxicity. Patients also undergo collection of blood, urine, stool, rectal swab samples, and rectal biopsies throughout the trial.
  Interventions: Drug: Aspirin; Procedure: Biospecimen Collection; Other: Questionnaire Administration; Procedure: Rectal Biopsy
- Arm II (aspirin, placebo) (Experimental): Patients receive aspirin PO daily at weeks 1-3 and 7-9 and placebo PO daily at weeks 4-6 and 10-12 in the absence of unacceptable toxicity. Patients also undergo collection of blood, urine, stool, rectal swab samples, and rectal biopsies throughout the trial.
  Interventions: Drug: Aspirin; Procedure: Biospecimen Collection; Other: Placebo Administration; Other: Questionnaire Administration; Procedure: Rectal Biopsy
- Arm III (placebo) (Placebo Comparator): Patients receive placebo PO daily for 12 weeks in the absence of unacceptable toxicity. Patients also undergo collection of blood, urine, stool, rectal swab samples, and rectal biopsies throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Placebo Administration; Other: Questionnaire Administration; Procedure: Rectal Biopsy

INTERVENTIONS:
Drug: Aspirin — Given PO
  Other Names: Acetylsalicylic Acid; ASA; Aspergum; Ecotrin; Empirin; Entericin; Extren; Measurin
  Arms: Arm I (aspirin); Arm II (aspirin, placebo)
Procedure: Biospecimen Collection — Undergo collection of blood, urine, stool, and rectal swab samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Placebo Administration — Given PO
  Arms: Arm II (aspirin, placebo); Arm III (placebo)
Other: Questionnaire Administration — Ancillary studies
Procedure: Rectal Biopsy — Undergo rectal biopsy
  Other Names: Biopsy of Rectum

SUMMARY:
This phase IIa trial studies how well aspirin works in preventing colorectal cancer in patients with colorectal adenoma. Aspirin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To test for the equivalency of the two aspirin schedules.

SECONDARY OBJECTIVES:

I. To evaluate the effects of aspirin treatments on:

Ia. The ratio of cell proliferation (Ki-67)/apoptosis (TUNEL) in rectal biopsies; Ib. The ratio of cell proliferation (Ki-67)/necroptosis (pMLKL) in rectal biopsies; Ic. Fecal occult blood test (measures of adverse events) as measured by stool samples.

EXPLORATORY OBJECTIVES:

I. To evaluate the effects of aspirin treatments on:

Ia. Cyclooxygenase-2 (COX-2) in rectal biopsies; Ib. Bcl-2-like protein 4 (BAX) in rectal biopsies; Ic. Transient receptor potential cation channel subfamily M member (7TRPM7) in rectal biopsies; Id. Joint index of COX-2 with TRPM7 expression in rectal biopsies; Ie. Joint index of TRPM7 with BAX in rectal biopsies; If. Methylation assays using the MethylationEPIC BeadChip to identify methylation biomarkers in genes (i.e. CDKN2A [cell cycle regulation], MGMT [deoxyribonucleic acid (DNA) repair], DAPK1 [apoptosis], CDH1 [cell invasion], WNT16 [Wnt pathway] and RASSF1 [RAS signaling]) involved in colorectal carcinogenesis, and other epigenome-wide methylation biomarkers as measured in rectal biopsies; Ig. Metagenomics analysis to measure abundance of Escherichia coli (E. coli) and Fusobacterium and other microbiota in rectal swabs.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive aspirin orally (PO) daily for 12 weeks in the absence of unacceptable toxicity. Patients also undergo collection of blood, urine, stool, rectal swab samples, and rectal biopsies throughout the trial.

ARM II: Patients receive aspirin PO daily at weeks 1-3 and 7-9 and placebo PO daily at weeks 4-6 and 10-12 in the absence of unacceptable toxicity. Patients also undergo collection of blood, urine, stool, rectal swab samples, and rectal biopsies throughout the trial.

ARM III: Patients receive placebo PO daily for 12 weeks in the absence of unacceptable toxicity. Patients also undergo collection of blood, urine, stool, rectal swab samples, and rectal biopsies throughout the trial.

After completion of study, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal adenoma of any grade
* Age >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of aspirin in participants < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 150,000/microliter
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional ULN
* Creatinine =< 1.5 x institutional ULN
* Blood hemoglobin >= 12.0 g/dL
* Alkaline phosphatase =< 1.5 x institutional ULN
* Blood urea nitrogen (BUN) =< 40 mg/dL
* Estimated glomerular filtration rate (eGFR) >= 45 mL/min
* Negative fecal occult blood test
* The effects of aspirin on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Current (within three weeks of randomization) or planned use during the study intervention of the following:

  * Aspirin, other nonsteroidal anti-inflammatory drugs (NSAIDs), or COX-2 inhibitors
  * Anticoagulants, anti-platelet agents, or corticosteroids
  * Gingko
  * Ethanol consumption > 1 standard drinks/day for women, or > 2 standard drinks/day for men
  * Methotrexate (MTX)
  * Study participants will be instructed to use Tylenol or some other non-excluded agent to treat common ailments (i.e. headache/minor aches and pains)
* History of

  * Any invasive malignancy within the past 2 years, with the exception of non-melanoma skin cancer
  * Chronic renal diseases or liver cirrhosis
  * Diseases such as anemia, peptic ulcer, gastrointestinal bleeding, active colitis and inflammatory bowel disease
  * Hemorrhagic stroke or uncontrolled hypertension
* Participants may not be receiving any other investigational agents
* History of allergic reactions or intolerance attributed to aspirin or compounds of similar chemical or biologic composition
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements
* Women who are pregnant or breastfeeding; pregnant women are excluded from this study because aspirin has the potential for abortifacient effects; because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with aspirin, breastfeeding should be discontinued if the mother is treated with aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-12-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Qi Dai, Principal Investigator — Northwestern University
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 81 participants were randomized. 70 out of the 81 started study agent.
Period: Overall Study
Arm/Group | Arm I (Aspirin) | Arm II (Aspirin, Placebo) | Arm III (Placebo)
Started | 29 | 33 | 8
Completed | 19 | 28 | 6
Not Completed | 10 | 5 | 2
Not completed — Withdrawal by Subject | 6 | 3 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: 81 participants were randomized. 70 out of the 81 started study agent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Aspirin) | Arm II (Aspirin, Placebo) | Arm III (Placebo) | Total
Number analyzed (Participants) | 36 | 36 | 9 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8) | 60 (6) | 57 (6) | 60 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 5 | 43
  Male | 19 | 15 | 4 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 35 | 36 | 9 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 0 | 9
  White | 32 | 31 | 9 | 72
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 9 | 81

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Cell Proliferation to Apoptosis Biomarkers (Ki67 Index and BAX Index)
Description: Change in the ratio of proliferation to apoptosis biomarkers (Ki67 density index: BAX density index, measured continuously after IHC staining) in colorectal mucosa of compliant participants
Time Frame: Baseline to end of intervention up to 12 weeks
Population: Participants with pre and post intervention samples available.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Arm I (Aspirin) | Arm II (Aspirin, Placebo) | Arm III (Placebo)
Number analyzed (Participants) | 14 | 23 | 4
ratio | -0.11 [-0.26 to 1.26] | 0.00 [-0.42 to 0.92] | -0.23 [-0.32 to -0.03]

2. Secondary Outcome: Ratio of Cell Proliferation (Ki-67)/Apoptosis (TdT-mediated dUTP Nick End Labeling [TUNEL]) in Rectal Biopsies
Description: Change in the ratio of proliferation to apoptosis biomarkers (Ki67 density index: TUNEL density index, measured continuously after IHC staining) in colorectal mucosa of compliant participants.
Time Frame: Baseline to end of intervention up to 12 weeks
Population: Participants with pre and post intervention samples available.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Arm I (Aspirin) | Arm II (Aspirin, Placebo) | Arm III (Placebo)
Number analyzed (Participants) | 14 | 23 | 4
ratio | -1.27 [-1.66 to 0.99] | 0.63 [-0.20 to 1.78] | -0.70 [-2.32 to 0.71]

3. Secondary Outcome: Ratio of Cell Proliferation (Ki-67)/Necroptosis (MLKL) in Rectal Biopsies
Description: Change in the ratio of proliferation to necroptosis biomarkers (Ki67 density index: pMLKLdensity index, measured continuously after IHC staining) in colorectal mucosa of compliant participants
Time Frame: Baseline to end of intervention up to 12 weeks
Population: Participants with pre and post intervention samples available.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Arm I (Aspirin) | Arm II (Aspirin, Placebo) | Arm III (Placebo)
Number analyzed (Participants) | 14 | 23 | 4
ratio | 0.58 [-0.84 to 0.79] | -0.02 [-0.53 to 0.39] | -0.32 [-1.39 to 0.77]

4. Secondary Outcome: Fecal Occult Blood Test (Measures of Adverse Events) as Measured by Stool Samples
Description: The number of participants who started intervention and had a positive fecal occult blood test result
Time Frame: Baseline to end of intervention up to 12 weeks.
Population: Participants with pre and post intervention samples available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Aspirin) | Arm II (Aspirin, Placebo) | Arm III (Placebo)
Number analyzed (Participants) | 20 | 30 | 7
Participants | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: AEs collected from the time of first dose of aspirin or placebo, through 40 days post-intervention.
Description: All participants will be evaluable for toxicity from the time of their first dose of aspirin or placebo
Arm/Group | Arm I (Aspirin) | Arm II (Aspirin, Placebo) | Arm III (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/33 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/33 | 1/8
Other Adverse Events (participants affected / at risk) | 7/29 | 9/33 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Aspirin) (N=29) | Arm II (Aspirin, Placebo) (N=33) | Arm III (Placebo) (N=8)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Kidney Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Aspirin) (N=29) | Arm II (Aspirin, Placebo) (N=33) | Arm III (Placebo) (N=8)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) — Blood in stool; Blood during bowel movement
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Abscess left axilla
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) — Sprained wrist; Small cut on head; Rectal sensitivity after biopsy
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT02965703/Prot_SAP_001.pdf